CLINICAL TRIAL: NCT02355613
Title: Comparative Evaluation of Two Different Radiosurgery Modalities in Brain Metastatic Patients From Several Solid Tumors
Brief Title: Comparative Evaluation of Two Different Radiosurgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, MD, Istituto Clinico Humanitas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1268
Record Dates: First submitted 2015-01-13; First posted 2015-02-04 (Estimated); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Metastases to Brain
Keywords: Radiosurgery, brain, metastases
MeSH Terms: conditions — Brain Neoplasms; Neoplasm Metastasis | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiosurgery with Gamma Knife Perfexion (Active Comparator): A single dose of 24 Gy at 50% isodose will be prescribed at metastases with diameter ≤ 20 mm, while a dose of 20 Gy at 50% isodose will be prescribed for metastases with diameter 21-30 mm
  Interventions: Radiation: Radiosurgery with Gamma Knife Perfexion
- Linac-based Radiosurgery with EDGE (Active Comparator): A single dose of 24 Gy will be prescribed at mean dose to PTV at metastases with diameter ≤ 20 mm, while a dose of 20 Gy will be prescribed for metastases with diameter 21-30 mm
  Interventions: Radiation: Linac-based Radiosurgery with EDGE

INTERVENTIONS:
Radiation: Radiosurgery with Gamma Knife Perfexion — Gamma Knife Radiosurgery is a very precise form of therapeutic radiology. Even though it is called surgery, a Gamma Knife procedure does not involve actual surgery but it uses 192 isocentric beams of highly-focused gamma rays (60-Co) to treat small to medium size lesions. Minimum beam size is 4 mm. This procedure is frame based.
  Arms: Radiosurgery with Gamma Knife Perfexion
Radiation: Linac-based Radiosurgery with EDGE — EDGE linear accelerator from Varian (Varian, Palo Alto, USA) is a C-arm machine specifically developed for radiosurgery frameless treatment. The characteristics of this linac are a high level of precision and the possibility to include multiple positioning systems for stereotactical treatments, among which Cone Beam CT (CBCT), the Optical Surface Monitoring System (OSMS), and Calypso.
  Arms: Linac-based Radiosurgery with EDGE

SUMMARY:
Randomized double arm phase III study to evaluate feasibility and safety of Gamma Knife radiosurgery and Linac Based (Edge) radiosurgery in brain metastatic patients

DETAILED DESCRIPTION:
This is a prospective double arm phase III study to evaluate cerebral side effects following radiosurgery delivered by Gamma Knife Perfexion and Linac Based EDGE. In particular our primary objective is to evaluate rate of symptomatic radionecrosis from the two different modalities of radiosurgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 85 years
* 1 - 4 brain metastases
* Karnofsky performance status (KPS) ≥70
* RPA 1 or 2
* Histopathologically confirmation of primary solid tumor
* Estimated survival ≥ 3 months as GPA score
* Written informed consent

Exclusion Criteria:

* Prior WBRT
* Age > 85 years
* KPS < 70
* RPA 3
* Diagnosis of small cell lung cancer (SCLC) or Lymphoproliferative disease
* Use of Avastin for at least 2 months after radiosurgery
* Pregnant women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2014-12-15 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
Incidence of symptomatic radionecrosis | two years

SECONDARY OUTCOMES:
Local Control of Brain Metastases | two years
Disease Free survival | two years
Overall survival | two years

CONTACTS AND LOCATIONS:
Overall Officials: Marta Scorsetti, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, MI, Italy

REFERENCES:
- [Derived] Scorsetti M, Navarria P, Cozzi L, Clerici E, Bellu L, Franceschini D, Marzo AM, Franzese C, Torri V, Reggiori G, Lobefalo F, Raspagliesi L, Attuati L, Pessina F, Franzini A, Picozzi P, Tomatis S. Radiosurgery of limited brain metastases from primary solid tumor: results of the randomized phase III trial (NCT02355613) comparing treatments executed with a specialized or a C-arm linac-based platform. Radiat Oncol. 2023 Feb 7;18(1):28. doi: 10.1186/s13014-023-02216-5. PMID 36750848